CLINICAL TRIAL: NCT06562959
Title: Effect of Integrating Auricular Acupressure and Fluid Restriction Program on Salivary Flow Rate and Fluid Control Adherence Among Children Undergoing Haemodialysis
Brief Title: Auricular Acupressure and Fluid Restriction Program on Salivary Flow and Fluid Adherence in Children on Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, Assisstant Profesor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AU-20-4-226-IRB00013620
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hemodialysis Complication
Keywords: Acupressure; Auricular; Fluid Control; Haemodialysis; Salivary Excretion; Therapeutic Adherence and Compliance
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The fluid restriction program included (a) General small-group discussion sessions, (b) individualized consultations, and (c) follow-up sessions.
  Interventions: Behavioral: Fluid Restriction Program
- Study Group (Experimental): The intervention bundle, the fluid restriction program, and auricular acupressure were received at four appointments: Shenmen, Kidney Concha, Point Zero, and Upper Tragus.
  Interventions: Other: Intervention Bundle (Fluid Restriction Program and Auricular Acupressure

INTERVENTIONS:
Behavioral: Fluid Restriction Program — In order to design the fluid restriction program content (booklet). The fluid restriction program included (a) General small-group discussion sessions, (b) individualized consultations, and (c) follow-up sessions. In the group discussion sessions, children in both the study and control groups were divided into subgroups (6 participants per each). In the group discussion sessions, children in both the study and control groups were divided into subgroups. The sessions were conducted in the meeting room of the Hemodialysis unit lasts for 45 minutes. In the Individualized Consultations, children then were provided tailored, age-appropriate education. The researchers also arranged for regular follow-up for one months.
  Arms: Control Group
Other: Intervention Bundle (Fluid Restriction Program and Auricular Acupressure — the study group received the Fluid Restriction Program and Auricular Acupressure in four acupoints namely, Shenmen, Kidney Concha, Point Zero and Upper Tragus. The researcher's finger gently pressed on each determined acupoints in a circular movement with a clockwise direction for three minutes.
  Arms: Study Group

SUMMARY:
This study aims to evaluate the effects of auricular acupressure on salivary flow rate and fluid restriction adherence among children undergoing Hemodialysis .

Hypothesis Children undergoing Hemodialysis who receive both auricular acupressure and fluid restriction program exhibit better salivary flow rate and fluid control adherence than those who receive fluid restriction program only.

DETAILED DESCRIPTION:
A non-randomized control trial was conducted at the Hemodialysis Unit in the Alexandria University Children's Hospital. A convenient sample of 60 children undergoing Hemodialysis was randomly assigned to two parallel groups. Both groups received the fluid restriction program in three types of sessions: general small-group discussion, individualized consultations, and follow-up. The study group also received auricular acupressure on four acupoints: Shenmen, Kidney Concha, Point Zero, and Upper Tragus.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 6 to 18 years
* Receiving hemodialysis for at least one month

Exclusion Criteria:

* Diabetes Mellitus
* Heart Diseases
* Autoimmune Disorders Such as Sjogren's Syndrome

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-03 (Actual)

PRIMARY OUTCOMES:
Salivary Flow Visual Analogue Scale | After one month
  This tool used to evaluate the salivary flow assessment. It consisted of 8 validated items measuring two main dimensions of salivary flow. The first dimension assessing the impaired oral functions due to the sensation of dry mouth as indicated by having difficulty in swallowing or speaking. While the second dimension evaluating the dryness of oral mucosa (lips, mouth, tongue, or throat). Additionally, children were asked two global questions regarding salivary quantity and thirsty level. In each item, children's responses were rated on a 100-mm horizontal numeric scale ranged from No (0) to very dry (100).

SECONDARY OUTCOMES:
Fluid Control in Hemodialysis Patients Scale | After one month
  This scale consisted of 24 items to evaluate the knowledge, behavior and attitude toward fluid restriction among patients undergoing hemodialysis. These items measure patients' compliance with fluid control.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Taha, Professor, Study Director — Alexandria University
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozen N, Cinar FI, Askin D, Mut D, Turker T. Nonadherence in Hemodialysis Patients and Related Factors: A Multicenter Study. J Nurs Res. 2019 Aug;27(4):e36. doi: 10.1097/jnr.0000000000000309. PMID 30720548
- [Background] Ahrari S, Moshki M, Bahrami M. The Relationship Between Social Support and Adherence of Dietary and Fluids Restrictions among Hemodialysis Patients in Iran. J Caring Sci. 2014 Feb 27;3(1):11-9. doi: 10.5681/jcs.2014.002. eCollection 2014 Mar. PMID 25276744
- [Background] Beerendrakumar N, Ramamoorthy L, Haridasan S. Dietary and Fluid Regime Adherence in Chronic Kidney Disease Patients. J Caring Sci. 2018 Mar 1;7(1):17-20. doi: 10.15171/jcs.2018.003. eCollection 2018 Mar. PMID 29637052
- [Background] Dembowska E, Jaron A, Gabrysz-Trybek E, Bladowska J, Trybek G. Oral Mucosa Status in Patients with End-Stage Chronic Kidney Disease Undergoing Hemodialysis. Int J Environ Res Public Health. 2023 Jan 2;20(1):835. doi: 10.3390/ijerph20010835. PMID 36613157
- [Background] Griva K, Nandakumar M, Ng JH, Lam KFY, McBain H, Newman SP. Hemodialysis Self-management Intervention Randomized Trial (HED-SMART): A Practical Low-Intensity Intervention to Improve Adherence and Clinical Markers in Patients Receiving Hemodialysis. Am J Kidney Dis. 2018 Mar;71(3):371-381. doi: 10.1053/j.ajkd.2017.09.014. Epub 2017 Dec 1. PMID 29198641
- [Background] Chang A, Chung Y, Kang M. Effects of the Combination of Auricular Acupressure and a Fluid-Restriction Adherence Program on Salivary Flow Rate, Xerostomia, Fluid Control, Interdialytic Weight Gain, and Diet-Related Quality of Life in Patients Undergoing Hemodialysis. Int J Environ Res Public Health. 2021 Oct 7;18(19):10520. doi: 10.3390/ijerph181910520. PMID 34639819
- [Derived] Rashwan ZI, Abdellah MMM, Moursi F, Ismail EMAE. Effect of bundling auricular acupressure and fluid restriction program on salivary flow rate and fluid control adherence among children undergoing hemodialysis: a randomized control trial. BMC Nurs. 2025 Jul 1;24(1):796. doi: 10.1186/s12912-025-03433-x. PMID 40597251